CLINICAL TRIAL: NCT02038166
Title: Chloride Secretagogues for Acquired CFTR Dysfunction in Chronic Rhinosinusitis (NPD Protocol)
Brief Title: Nasal Potential Difference (NPD) Protocol in Chronic Rhinosinusitis
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brad Woodworth, MD, Associate Professor of Surgery, University of Alabama at Birmingham
Other Study IDs: IRB-100930005; 1K08HL107142-01 (NIH)
Record Dates: First submitted 2014-01-09; First posted 2014-01-16 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
The purpose of this study is to determine if acquired (partial) Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) deficiency contributes substantially to the pathogenic mechanisms underlying Chronic Rhinosinusitis (CRS), creating a localized environment that impairs mucociliary clearance (MCC).

DETAILED DESCRIPTION:
Nasal Potential Difference (NPD) measurements will be conducted on participants. The NPD measurement, is a bioelectric assay of CFTR-dependent ion transport that has been used in a variety of protocols designed to detect CFTR function. A 4-Step protocol will be utilized. The nasal cavities will be perfused in a step-wise fashion with the following solutions: 1) Ringer's solution, 2) Ringer's solution + amiloride 100μM, 3) Low-Cl--containing solution, and 4) Low-Cl- + isoproterenol (10 µM). The potential difference will be monitored in nasal epithelium in comparison to an agar filled reference butterfly electrode placed in the volar aspect of the forearm, and connected via a calomel cell to a high impedance voltmeter.

Following placement of the subcutaneous reference bridge, the nasal probe will be secured 1-3 cm within the inferior meatus and secured in position at the most polarizing position. Each nare will then be sequentially perfused with Ringer solution. All nasal potential difference tracings will be scored independently by a single reviewer.

The investigator and an internal committee comprised of Gregory Fleming James Associate Scientists will oversee the safety of the study. Our internal committee is a multidisciplinary group consisting of physician and subspecialists who, collectively, have experience in treatment patients with cystic fibrosis and other airway disease in the conduct of randomized clinical trials. The primary responsibility of this committee is to protect the safety and welfare of subjects consenting to the investigator's procurement of remnant tissue during endoscopic sinus procedure. Members are responsible for reviewing procedural conduct, including acquisition of consents and materials, to protect patient well-being. An interim data safety review will be conducted on a yearly basis. The committee will consist of at least 3 members with clinical trials experience in airway diseases. During annual review, issues relating to the safety and process for acquiring human tissues will be reviewed. Summary reports from each annual meeting will be prepared and will address concerns about the procurement of tissue or any other information deemed pertinent to the review.

ELIGIBILITY:
The patient eligibility criteria are designed to limit enrollment to healthy individuals and patients who clearly have CRS based on Sinus and Allergy health partnership criteria, but who are sufficiently well (both in terms of CRS and in terms of concomitant illness, such as asthma) to safely participate in study procedures and provide interpretable results.

Inclusion Criteria:

a. Patients with CRS will be diagnosed according to Sinus and Allergy Health Partnership symptom-based and objective criteria as follows: i. Duration of disease is qualified by continuous symptoms (≥ 2 major factors or at least 1 major factor & 2 minor symptoms; Table 2) for ≥ 12 consecutive weeks or ≥ 12 weeks of physical findings. ii. One of these signs of inflammation must be present and identified in association with ongoing symptoms.

1. Discolored nasal drainage arising from the nasal passages, nasal polyps, or polypoid swelling as identified on physical examination with nasal endoscopy.
2. Edema or erythema of the middle meatus or ethmoid bulla
3. Generalized or localized erythema or edema. If it does not involve the middle meatus or ethmoid bulla, CT scan is performed to confirm a diagnosis.
4. The CT scan must demonstrate isolated or diffuse mucosal thickening, bone changes, air-fluid levels. b. Age ≥ 19 years and Weight ≥ 50 kg c. Ability to perform NPD testing d. Negative pregnancy test (for females of childbearing potential) e. Written informed consent

Exclusion Criteria:

1. Acute illness within 2 weeks before start of study treatment.
2. History of major asthma attack within 2 months prior to start of study treatment.
3. Change in intranasal medications (including use of corticosteroids, cromolyn, atrovent, phenylephrine, or oxymetazoline) within 14 days prior to start of study treatment.
4. Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test.
5. Hemoglobin <10 gm/dL and Serum albumin <2.5 g/dL.
6. Abnormal liver function (serum ALT, AST, alkaline phosphatase, or total bilirubin >2 times upper limit of normal).
7. Abnormal renal function (serum creatinine >1.5 times upper limit of normal).
8. Pregnancy or breast feeding.
9. History of solid organ or hematological transplantation
10. History of autoimmune or granulomatous disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to UAB for evaluation of CRS
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Measurable Difference in CFTR function | One Year
  A >-5 mV increase in total chloride secretion (change in NPD following nominal Cl- solution + amiloride + isoproterenol) is typically designated as evidence of measurable difference in CFTR function. Results of NPD measurements between CRS patients and healthy controls will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Woodworth, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States